CLINICAL TRIAL: NCT07108543
Title: Antegrade Versus Retrograde Cross K-Wire In Distal Radius Fracture; A Comparative Study
Brief Title: Antegrade Versus Retrograde Cross K-Wire In Distal Radius Fracture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Montasser Talaat Omar, resident orthopeadics sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25--24MS
Record Dates: First submitted 2025-07-30; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial using a parallel assignment model. Participants will be randomly assigned to one of two groups: Group A will undergo cross K-wire fixation using the antegrade technique, and Group B will undergo the retrograde technique. Outcomes will be compared between the two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Title: Antegrade K-wire Fixation (Experimental): participants in this group will undergo antegrade percutaneous cross K-wire fixation for distal radius fractures. K-wires will be inserted from proximal to distal direction under fluoroscopic guidance, following closed reduction
  Interventions: Procedure: Antegrade versus retrograde cross k-wire
- Arm 2 Title: Retrograde K-wire Fixation (Experimental): Participants in this group will undergo retrograde percutaneous cross K-wire fixation for distal radius fractures. K-wires will be inserted from distal to proximal direction under fluoroscopic guidance, following closed reduction
  Interventions: Procedure: Antegrade versus retrograde cross k-wire

INTERVENTIONS:
Procedure: Antegrade versus retrograde cross k-wire — > Closed reduction of distal radius fracture followed by percutaneous insertion of two or more K-wires in an antegrade direction (from proximal to distal), crossing the fracture site under fluoroscopic guidance. The wires are introduced from the radial metaphysis and directed distally to stabilize the fracture.

SUMMARY:
This study aims to compare the clinical and radiological outcomes of distal radius fractures treated with cross K-wire fixation using the antegrade versus retrograde technique. Adult patients with extra-articular distal radius fractures will be randomly assigned to one of the two surgical approaches. The primary outcomes include fracture stability, functional recovery, and complication rates. The study is designed as a prospective, randomized controlled trial conducted at sohag university

ELIGIBILITY:
Inclusion Criteria:

Patients with extra-articular distal radius fractures. Fractures classified as Frykmann type 1 and type 2. Patients aged 18 years and above.

Exclusion Criteria:

* Skeletally immature patient.
* Intra-articular distal radius fractures.
* Communited fractures.
* Open fractures or fractures with neurovascular compromise.
* Patients with fractures requiring surgical interventions other than K-wire fixation.
* Patients with a history of infection or other conditions impair wound healing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Radiological union of distal radius fracture | At 6 weeks, 3 months, and 6 months postoperatively
  Radiographic healing will be assessed using standard X-rays to evaluate union status. Radiographs will be reviewed for signs of cortical continuity and absence of fracture lines

SECONDARY OUTCOMES:
Functional outcome using DASH score | At 6 weeks, 3 months, and 6 months postoperatively
  Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will be used to assess upper limb function
Pain level using Visual Analog Scale (VAS) | At 1 week, 6 weeks, 3 months, and 6 months postoperatively
  Pain will be evaluated using the Visual Analog Scale (0-10), with 0 indicating no pain and 10 indicating worst pain